CLINICAL TRIAL: NCT01684644
Title: Parent Training for Preschool ADHD: A Randomised Controlled, Multicentre Effectiveness Trial of the New Forest Parenting Programme in a Clinical Sample of Danish Children
Brief Title: A Controlled Study of Parent Training in the Treatment of ADHD in Young Children
Acronym: D'SNAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); TrygFonden, Denmark (Industry); Sygekassernes Helsefond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7-10-1294; 7-10-1294 (Other Grant/Funding Number: 7-10-1294)
Record Dates: First submitted 2012-09-04; First posted 2012-09-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Parent Training; RCT; Preschool
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Forest Parenting Programme (Experimental): The New Forest Parenting Programme is a parent training programme specifically developed to treat ADHD in preschool children. The programme is delivered as an 8 week intervention for individual parents and their child.
  Interventions: Behavioral: New Forest Parenting Programme
- Treatment as Usual (Other): Treatment as usual for preschool ADHD consists of psychoeducation groups for parents.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: New Forest Parenting Programme
  Arms: New Forest Parenting Programme
Behavioral: Treatment as usual
  Other Names: Psychoeducation in groups for parents of young children diagnosed with ADHD
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to investigate the effectiveness of parent training in the treatment of ADHD in young children (ages 3-7) referred to Danish child mental health services. Medication is not recommended as first-line treatment for young children with ADHD. Parent training is recommended, but has not been formally introduced or established in Denmark. The study will investigate the effectiveness of a parent training programme specifically developed to target ADHD symptoms in young children; The New Forest Parenting Programme, against Treatment as Usual for children diagnosed with ADHD at two different child mental health clinics in Denmark.

DETAILED DESCRIPTION:
Description: A study to: 1) Address the need for non-pharmacological treatment in young children with ADHD and 2) Address the need for the development of evidence-based psychosocial treatment interventions in Danish child mental health services, through the implementation of the New Forest Parenting Programme (NFPP).

Rationale: ADHD is a neuro-developmental disorder with symptoms frequently occurring in early childhood. ADHD is associated with long-term personal, psychosocial sequalae. ADHD presents a considerable societal cost burden, both for mental health services, but also in areas such as education, employment, the criminal justice system. Pharmacological treatment of preschool ADHD is not recommended as first-line treatment, due to a number of reasons, including lack of evidence for efficacy, parental concerns, side effects on growth rates, and the unknown long-term implications for the developing brain. Effective psychosocial treatments for ADHD are therefore of central public priority generally, and for child mental health services, specifically. Currently, psychosocial interventions for ADHD in pre-school children in Danish Child and Adolescent Mental Health Services (CAMHS) are not well described or systematically developed. There is a pressing need to develop evidence-based psycho-social treatments for young children with ADHD in Danish CAMHS.

Design: The study will be a randomised controlled multi-centre effectiveness trial comparing NFPP intervention to a Treatment as Usual control group. The trial will recruit 200 preschool children (aged 3-6) with a diagnosis of ADHD from two Danish outpatient child mental health service sites. Participants will be randomised to either 1) NFPP over a period of 8 weeks or 2) a control group receiving Treatment as Usual (TAU). Outcome: The primary outcome measure will be child ADHD symptoms. Secondary outcomes include parental wellbeing, child quality of life, parent-child interactions. Measures will be collected at three time points to track changes in outcome: T1: Before start of intervention or TAU condition. T2: Directly after the intervention or TAU and T3: 6 month follow-up after T1 for both arms of the trial. The study will perform exploratory moderator and mediator analyses.

Expertise: The study receives external consultation from an international expert team for the planning, execution, NFPP training and supervision. The team consists of research and clinical experts in the treatment and evaluation of interventions for preschool ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of ADHD, as measured by the DAWBA
2. Participants first language must be Danish

Exclusion Criteria:

1. Children with intellectual disabilities (i.e. IQ < 70), Autism Spectrum Disorders.
2. Severe parental psychiatric disorder
3. Severe social adversity, as defined by social services involvement due to suspicions of or detected neglect.
4. Child receiving medication or other treatment for ADHD symptoms

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 164 (Actual)
Dates: Start 2012-09; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale IV-Preschool Version | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  A screening instrument for the symptoms of AD/HD in the preschool population.

SECONDARY OUTCOMES:
Preschool ADHD-RS (Teacher completed) 18 items | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  screening instrument for the symptoms of AD/HD in the preschool population.
Strength and Difficulties Questionnaire (parent version) | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  A brief measure of prosocial behaviour and and psychopathology of 3-16 year olds that can be completed by parents
Strength and Difficulties Questionnaire (teacher completed) | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  A brief measure of prosocial behaviour and and psychopathology of 3-16 year olds that can be completed by teachers
Child solo play - observation measure - | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  Observation measure: Index of Attention scale assessed from 'time on task'/no. of switches in activity' with high scores representing more attention and less switching
Child Health Questionnaire (CHQ-28) | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  Quality of life measure
Family Strain Index 6 items | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  Short screening instrument for the detection of family strain

OTHER OUTCOMES:
Parental report on somatic complaints in preschool children | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  Parental report on somatic complaints in preschool children (Domenech-Llaberia et al., 2004)
6. The Adult ADHD self-report scale (ASRS-V1.1) 18 items The Adult ADHD self-report scale (ASRS-V1.1) 18 items | T1 (Baseline)
  Adult ADHD screening instrument
Parent sense of competence scale (PSOC) (17 items) | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  Instrument to assess perceived sense of parenting competence
Maternal expressed emotion - 5 min speech sample. | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  A 5-min speech sample obtained from mothers, rated over 6 scales with an overall high score indicating a negative influence on the child.
GIPCI (Jigsaw/Tidy up/Freeplay) observation measure | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  GIPCI (Jigsaw/Tidy up/Freeplay) observation measure of parent child interaction with global ratings (0-5) for parent and child behaviours
General Health Questionnaire (12 item) | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)
  Screening instrument to detect psychiatric disorders in adults
Neuropsychological test battery | T1 (at baseline), T2 (twelve weeks from T1)
  Working memory (verbal and visuospatial) measured by Word span Forward and Backward as well as using Finger Windows Forward and Backward.
  Inhibition measured using a modified four picture pairs Stroop Task as well as the Head-Toes-Knees-Shoulders task.
  Flexibility measured using the Switching, Inhibition, and Flexibility Task as well as the Trails-P.
  Delay-related behavior measured with the Cookie Delay Task and the Teddy Delay Task
  Simple information processing time measured using the Fish task.
  In addition, video recordings of the neuropsychological evaluation will be coded and analyzed (private speech and behavior) after the test session
Behavior Rating Inventory of Executive Function - Preschool Version [BRIEF-P] | T1 (at baseline), T2 (twelve weeks from T1), T3 (6 months from T1)

CONTACTS AND LOCATIONS:
Overall Officials: Per Hove Thomsen, MD, Study Chair — Børne- og Ungdomspsykiatrisk Center-Risskov, Aarhus Universitetshospital, Skovagervej 2, 8240 Risskov, Denmark
Locations (1):
- Center for child and adolescent psychiatry, Risskov, Aarhus, Denmark

REFERENCES:
- [Derived] Larsen LB, Daley D, Lange AM, Sonuga-Barke E, Thomsen PH, Rask CU. Effect of Parent Training on Health-Related Quality of Life in Preschool Children With Attention-Deficit/Hyperactivity Disorder: A Secondary Analysis of Data From a Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2021 Jun;60(6):734-744.e3. doi: 10.1016/j.jaac.2020.04.014. Epub 2020 Jun 4. PMID 32505701
- [Derived] Lange AM, Daley D, Frydenberg M, Houmann T, Kristensen LJ, Rask C, Sonuga-Barke E, Sondergaard-Baden S, Udupi A, Thomsen PH. Parent Training for Preschool ADHD in Routine, Specialist Care: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2018 Aug;57(8):593-602. doi: 10.1016/j.jaac.2018.04.014. Epub 2018 Jun 18. PMID 30071980
- [Derived] Lange AM, Daley D, Frydenberg M, Rask CU, Sonuga-Barke E, Thomsen PH. The Effectiveness of Parent Training as a Treatment for Preschool Attention-Deficit/Hyperactivity Disorder: Study Protocol for a Randomized Controlled, Multicenter Trial of the New Forest Parenting Program in Everyday Clinical Practice. JMIR Res Protoc. 2016 Apr 13;5(2):e51. doi: 10.2196/resprot.5319. PMID 27076496